CLINICAL TRIAL: NCT04576104
Title: Surgical Window of Opportunity Study of Megestrol Acetate Compared With Megestrol Acetate and Metformin for Endometrial Intraepithelial Neoplasia
Brief Title: Megestrol Acetate Compared With Megestrol Acetate and Metformin to Prevent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2020-07529; NCI-2020-07529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI20-02-01 (Other: Northwestern University); NWU20-02-01 (Other: DCP); P30CA060553 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2020-10-03; First posted 2020-10-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Atypical Hyperplasia/Endometrioid Intraepithelial Neoplasia; Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Biopsy; Metformin; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (megestrol acetate) (Active Comparator): Prior to standard of care planned procedure, patients receive megestrol acetate PO BID for 21-35 days (up to and including the night before planned procedure) in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on the day of planned procedure.
  Interventions: Procedure: Biopsy Procedure; Drug: Megestrol Acetate; Other: Questionnaire Administration
- Arm II (megestrol acetate, metformin hydrochloride) (Experimental): Prior to standard of care planned procedure, patients receive megestrol acetate PO BID and metformin hydrochloride extended-release PO BID for 21-35 days (up to and including the night before planned procedure) in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on the day of planned procedure.
  Interventions: Procedure: Biopsy Procedure; Drug: Extended Release Metformin Hydrochloride; Drug: Megestrol Acetate; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Drug: Extended Release Metformin Hydrochloride — Given PO
  Other Names: ER Metformin Hydrochloride; Extended-release Metformin Hydrochloride; Glucophage XR; Glumetza; Metformin Hydrochloride Extended Release
  Arms: Arm II (megestrol acetate, metformin hydrochloride)
Drug: Megestrol Acetate — Given PO
  Other Names: 17-Hydroxy-6-methylpregna-4,6-diene-3,20-dione acetate; 17.alpha.-Acetoxy-6-methylpregna-4,6-diene-3,20-dione; 6-Dehydro-6-methyl-17.alpha.-acetoxyprogesterone; 6-Methyl-6-dehydro-17.alpha.-acetoxyprogesterone; BDH 1298; BDH-1298; Maygace; Megace; Megestat; Megestil; Niagestin; Ovaban; Pallace; SC 10363; SC-10363
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of megestrol acetate alone or in combination with metformin in preventing the progression of uterine pre-cancer (endometrial intraepithelial neoplasia) to endometrial cancer. Megestrol acetate is a drug used to block estrogen and suppress the effects of estrogen and androgens. It is the current non-surgical treatment of endometrial intraepithelial neoplasia. Metformin is a drug that has been found to have anti-cancer properties. Giving metformin and megestrol acetate together may decrease the growth of endometrial intraepithelial neoplasia in the uterus better than megestrol alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the change in endometrial cell proliferation, as measured by the percentage (%) of Ki-67 positive cells, in participants with endometrial intraepithelial neoplasia who undergo 4 weeks of treatment with megestrol acetate + metformin or megestrol acetate alone prior to planned procedure (hysterectomy) or progestin intrauterine device [IUD] placement).

SECONDARY OBJECTIVE:

I. To measure the changes in protein expression in the endometrial intraepithelial neoplasia lesion, using immunohistochemistry (i-vi) in subjects treated with megestrol acetate + metformin compared to those treated with megestrol acetate alone.

i. Estrogen receptor (ER) and progesterone receptor (PR) ii. PTEN/PAX2 expression iii. Markers of the PI3K-Akt-mTOR pathway (phosphor-acetyl-CoA carboxylase (ACC), p(Ser473)-Akt, phosphor-S6K, p4EBP1) iv. Markers of cell death (TUNEL, cleaved caspase-3) v. Markers of intratumoral insulin signaling (Phosphorylated insulin receptor (pIR) and insulin-like growth factor-1 receptor (total and phosphorylated IGF1R), vi. Mismatch repair (MMR) deficiency (baseline only).

EXPLORATORY OBJECTIVE:

I. To explore whether baseline Ki-67 expression and other clinical characteristics are associated with treatment response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Prior to standard of care planned procedure, patients receive megestrol acetate orally (PO) twice daily (BID) for 21-35 days (up to and including the night before planned procedure) in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on the day of planned procedure.

ARM II: Prior to standard of care planned procedure, patients receive megestrol acetate PO BID and metformin hydrochloride extended-release PO BID for 21-35 days (up to and including the night before planned procedure) in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on the day of planned procedure.

After completion of study treatment, patients are followed for up to 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with endometrial intraepithelial neoplasia (EIN) on an endometrial biopsy or dilation and curettage specimen will be eligible. Participants diagnosed with EIN bordering on, approaching or suspicious for endometrial adenocarcinoma are allowed. Participants can be diagnosed with EIN at any time in the three months prior to enrollment. Other commonly used pathologic terms for EIN, such as complex atypical hyperplasia and atypical hyperplasia will also be eligible
* Age >= 18 years-old. EIN is almost exclusively an adult condition. Because no dosing or adverse event (AE) data are currently available on the use of megestrol acetate in participants < 18 years of age, children and adolescents are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* If the participant is diabetic, blood glucose must be appropriately controlled as evidenced by a hemoglobin A1c of < 8.0 in the last three months prior to enrollment. If no A1c is available, it will be drawn with baseline laboratory parameters as is standard of care. For women who are diabetics who are on insulin, metformin can cause relative hypoglycemia. Women who are diabetic and receiving insulin will be allowed to participate, but will be asked to monitor their blood glucoses closely and alert the study team if persistent hypoglycemia is noted
* Must be a candidate and accepting of surgical management of EIN with planned hysterectomy or non-surgical treatment with a progestin IUD
* The effects of megestrol acetate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately. For metformin, published studies with metformin use during pregnancy have not reported a clear association with metformin and major birth defect or miscarriage risk. Metformin can increase the potential for unintended pregnancy in premenopausal women as therapy with metformin may result in ovulation in some anovulatory women
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current hormonal contraceptives or post-menopausal hormone replacement therapy, and uses of progestins (including progestin containing intrauterine device [IUD]) EXCEPT FOR:

  * Megestrol acetate up to and including 40 mg daily
  * Medroxyprogesterone acetate up to and including 10 mg daily
  * Norethindrone acetate up to and including 10 mg daily
  * Norethindrone up to and including 0.35 mg daily
  * Oral micronized progesterone up to and including 30 0mg daily These low potency and lower dose progestins are permitted provided they have been used for less than 8 weeks (56 days) prior to enrollment and were started after the pre-treatment biopsy (e.g. endometrial biopsy or dilation and curettage). Participants will discontinue these low potency and lower dose progestins at the time of enrollment NOTES: Vaginal estrogen use is permitted. Prior use of hormonal contraceptives or post-menopausal hormone therapy is allowed, provided that it was discontinued > 3 months from current EIN diagnosis.
* Current use of selective estrogen receptor modulators (SERMs) and aromatase inhibitors. Prior use of SERMs or aromatase inhibitors is allowed, provided that it was discontinued > 3 months from current EIN diagnosis
* Current use of metformin therapy (prior use of metformin therapy is allowed, provided that it was discontinued > 1 year from trial enrollment)
* Use of GLP-1 or dual GLP-1/GIP-1 receptor agonists within 6 weeks prior to the baseline diagnostic biopsy or randomization
* Participants receiving any other investigational agents within 30 days of enrollment or during this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or megestrol acetate
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because it requires hysterectomy or progestin IUD placement which is contraindicated in women who are pregnant and wish to continue the pregnancy. Additionally, megestrol acetate is a category D agent. Megestrol acetate may cause fetal harm when administered to a pregnant woman
* Women who are breastfeeding are excluded because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with megestrol acetate. Breastfeeding should be discontinued if the mother is treated with megestrol acetate
* Personal history of pulmonary embolism, thrombotic stroke, arterial thrombosis or deep vein thrombosis of the extremity or deep vein thrombosis
* Women who are diabetics on insulin will be eligible to participate but they will be required to check their blood sugar regularly. Patients who are unable to check their blood sugar will be excluded from participation
* Women who are diabetics taking sulfonylureas and meglitinides will be excluded
* Women with an alcohol use or abuse disorder due to increased risk of lactic acidosis with metformin
* Current use of dofetilide, ulipristal, or carbonic anhydrase inhibitors as well as drugs that reduce metformin clearance such as ranolazine, vandetanib, dolutegravir, or cimetidine
* Cancer survivors with evidence of active disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Ki-67 positive cells | Up to 42 days post planned procedure
  Will measure the change in endometrial cell proliferation, as measured by the percentage of Ki-67 positive cells, in subjects treated with megestrol acetate + metformin compared to those treated with megestrol acetate alone, in all evaluable participants, and following stratification by menopausal status, as well as use of low dose, low potency progestins (yes/no).

SECONDARY OUTCOMES:
Changes in protein expression | Baseline up to 42 days post planned procedure
  Measured by immunohistochemistry of samples in subjects treated with megestrol acetate + metformin compared to those treated with megestrol acetate alone. Additional analyses will be stratified for premenopausal and postmenopausal status, as well as use of low dose, low potency progestins (yes/no) to assess whether there are biologic differences in these two groups of women. i. Estrogen receptor and progesterone receptor; ii. PTEN/PAX2 expression; iii. Markers of the PI3K-Akt-mTOR pathway (phosphor-acetyl-CoA carboxylase, p(Ser473)-Akt, phosphor-S6K, p4EBP1);iv. Markers of cell death (TUNEL, cleaved caspase-3);v. Markers of intratumoral insulin signaling (Phosphorylated insulin receptor and insulin- like growth factor-1 receptor (total and phosphorylated IGF1R); vi. Mismatch repair deficiency (baseline only).

OTHER OUTCOMES:
Ki-67 expression | Baseline
  Will explore whether baseline Ki-67 expression and other clinical characteristics are associated with treatment response. Will measure differences in the changes of Ki-67 expression of samples in subjects treated with megestrol acetate + metformin compared to those treated with megestrol acetate alone based upon the following characteristics: Baseline Ki-67 expression, ribonucleic acid sequencing analysis, and clinical characteristics (body mass index, age, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm